CLINICAL TRIAL: NCT01314911
Title: A Randomized Double-Blind Study Comparing Oseltamivir Versus Placebo for the Treatment of Influenza in Low Risk Adults
Brief Title: Evaluating the Use of Oseltamivir for the Treatment of Influenza in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRC 004; 11-I-0031; IRC004
Record Dates: First submitted 2011-03-03; First posted 2011-03-15 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Influenza, Human
Keywords: H1N1; Complications; PCR; Seasonal Influenza; Viral Shedding
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oseltamivir (Experimental)
  Interventions: Drug: Oseltamivir
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oseltamivir — Subjects were prescribed Oseltamivir twice daily for 5 days, and each dose consisted of one capsule of Oseltamivir 75 mg.
  Arms: Oseltamivir
Drug: Placebo — Subjects were prescribed the matching placebo twice daily for 5 days, and each dose consisted of one capsule of placebo.
  Arms: Placebo

SUMMARY:
People who are infected with the influenza virus may develop respiratory illnesses, such as pneumonia, or other life-threatening complications. Currently, there are four antiviral medications that are used to treat influenza. This study will examine one of these medications, oseltamivir, to examine how it affects the shedding of influenza virus in infected people.

DETAILED DESCRIPTION:
Seasonal influenza is responsible for excess hospitalizations and, despite effective antivirals, causes significant morbidity and mortality (about 24,000 deaths each year in the United States alone). The influenza virus that emerged in 2009 (A/California/07/2009 H1N1) caused fewer deaths (12,000 flu-related deaths in the U.S.) but in contrast to seasonal flu, nearly 90% of the deaths with the 2009 H1N1 occurred among people younger than 65 years of age. Although there are four currently licensed anti-influenza medications (amantadine and rimantadine, oseltamivir, and zanamivir), previous studies have not demonstrated conclusively to what extent these medications affect influenza viral shedding. This study will evaluate whether oseltamivir modifies the viral shedding during the treatment of uncomplicated influenza in an adult population and also assess methods to detect viral replication in the upper respiratory tract.

Subjects who presented with an influenza-like illness without any risk factors for severe disease were screened for the study. Those with a confirmatory test for influenza (rapid antigen or polymerase chain reaction [PCR]) were randomized in a 1:1 manner to receive a blinded study treatment consisting of either the oseltamivir or placebo for 5 days. Clinical, virologic, and laboratory assessments on Days 1, 3, 7, and 28 were used for both safety and efficacy analysis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to initiation of any study procedures
* History of an influenza-like illness defined as:

  1) One or more respiratory symptom (cough, sore throat, or nasal symptoms)
* Onset of illness no more than 48 hours before screening, defined as when the participant experienced at least one respiratory symptom
* Willing to have samples stored
* Positive test for influenza (either rapid antigen or polymerase chain reaction [PCR]); randomization could proceed in cases of discrepant results (one positive and one negative)

Exclusion Criteria:

* Hospitalization at the time of screening
* Presence of a medical condition(s) that had been associated with increased risk of complications from influenza

  1. Aged 65 years of age or older
  2. Asthma
  3. Neurological and neuro-developmental conditions (including disorders of the brain, spinal cord, peripheral nerve, and muscle, such as cerebral palsy, epilepsy [seizure disorders], stroke, moderate to severe developmental delay, muscular dystrophy, or spinal cord injury)
  4. Chronic lung disease (such as chronic obstructive pulmonary disease [COPD] or cystic fibrosis)
  5. Heart disease (such as congenital heart disease, congestive heart failure, or coronary artery disease)
  6. Blood disorders
  7. Endocrine disorders (such as diabetes mellitus)
  8. Kidney disorders
  9. Liver disorders
  10. Metabolic disorders (such as inherited metabolic disorders or mitochondrial disorders)
  11. Weakened immune system due to disease or medication (such as people with HIV/AIDS or cancer, or use of chronic steroids or other medications causing immune suppression)
  12. Pregnant or 4 weeks postpartum
  13. Body mass index (BMI) greater than or equal to 40
* Breastfeeding
* Inability to take oral medication or a history of gastrointestinal malabsorption that would preclude the use of oral medication
* Received more than one dose of any antiviral influenza medication since onset of influenza symptoms
* Known end stage kidney dysfunction (e.g., creatinine clearance less than 30 mL/min)
* Known hypersensitivity to oseltamivir, peramivir, or zanamivir
* Received live attenuated influenza virus vaccine within 3 weeks prior to study entry
* Use of any investigational drug within 30 days or 5 half-lives (whichever was longer) prior to study entry
* Participated in other research protocols that required more than 100mL of blood to be drawn in a 4-week period that overlapped with this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 716 (Actual)
Dates: Start 2011-04; Primary Completion 2017-11-18 (Actual); Study Completion 2017-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Beigel, MD, Study Chair — Leidos Biomedical Research, Inc. in support of Clinical Research Section, LIR, NIAID, National Institutes of Health; Michael Ison, MD, MS, Study Chair — Division of Infectious Disease, Feinberg School of Medicine, Northwestern University
Locations (51):
- United States (44):
  - East Valley Family Physicians, Chandler, Arizona
  - WCCT Global, LLC, Costa Mesa, California
  - Paragon Rx Clinical, Garden Grove, California
  - University of Southern California, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Westlake Medical Research, Thousand Oaks, California
  - Advanced Rx Clinical Research Group, Westminster, California
  - University of Colorado, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Best Quality Research, Inc., Hialeah, Florida
  - Medical Consulting Center, Miami, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - University of Iowa, Iowa City, Iowa
  - Research Integrity, LLC, Owensboro, Kentucky
  - Horizon Research Group of Opelousas, LLC, Eunice, Louisiana
  - Michael Seep, MD; Centex Studies, Lake Charles, Louisiana
  - National Institutes of Health, Laboratory of Immunoregulation, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Skyline Medical Center, Elkhorn, Nebraska
  - Prairie Fields Family Medicine, Fremont, Nebraska
  - Southwest Family Physicians, Omaha, Nebraska
  - Clinical Research Advantage, Inc., Omaha, Nebraska
  - New Jersey Medical School, Newark, New Jersey
  - NYU School of Medicine, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Great Lakes Medical Research, Westfield, New York
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - University of Pennsylvania, Division of Infectious Disease, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Clinical Research Solutions, Franklin, Tennessee
  - Clinical Research Solutions, Jackson, Tennessee
  - Clinical Research Solutions, Nashville, Tennessee
  - Clinical Research Solutions, Smyrna, Tennessee
  - University of Texas Tech Amarillo, Amarillo, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Centex Studies, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Village Health Partners, Plano, Texas
  - Bandera Family Health Care, San Antonio, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
- Argentina (3):
  - Hospital General de Agudos J. M. Ramos Mejía, Buenos Aires
  - Hospital Municipal "Prof. Dr. Bernardo A. Houssay", Buenos Aires
  - Hospital Público Descentralizado Dr. Guillermo Rawson, Córdoba
- Thailand (4):
  - The Bamrasnaradura Infectious Diseases Institute, Nonthaburi, Changwat Nonthaburi
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok
  - Siriraj Hospital, Bangkok
  - Khon Kaen University (Department of Medicine), Khon Kaen

REFERENCES:
- [Background] Thompson WW, Shay DK, Weintraub E, Brammer L, Cox N, Anderson LJ, Fukuda K. Mortality associated with influenza and respiratory syncytial virus in the United States. JAMA. 2003 Jan 8;289(2):179-86. doi: 10.1001/jama.289.2.179. PMID 12517228
- [Background] Monto AS. Vaccines and antiviral drugs in pandemic preparedness. Emerg Infect Dis. 2006 Jan;12(1):55-60. doi: 10.3201/eid1201.051068. PMID 16494718
- [Derived] Beigel JH, Manosuthi W, Beeler J, Bao Y, Hoppers M, Ruxrungtham K, Beasley RL, Ison M, Avihingsanon A, Losso MH, Langlois N, Hoopes J, Lane HC, Holley HP, Myers CA, Hughes MD, Davey RT. Effect of Oral Oseltamivir on Virological Outcomes in Low-risk Adults With Influenza: A Randomized Clinical Trial. Clin Infect Dis. 2020 May 23;70(11):2317-2324. doi: 10.1093/cid/ciz634. PMID 31541242
- See also: The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009). — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with an influenza-like illness and diagnosed with influenza by rapid antigen or PCR were recruited at 42 sites from 3 countries: 3 from Argentina, 4 from Thailand and 35 from the U.S., between January 2012 to October 2017.
Pre-assignment Details: Seven hundred and sixteen subjects were enrolled per protocol (signed consent). Of these 716 subjects, three subjects were inadvertent enrollments, and one was a repeat enrollment of a subject who had been previously enrolled .One hundred fifty-four subjects were excluded during screening and did not participate in any other aspect of the trial.
Period: Overall Study
Arm/Group | Oseltamivir | Placebo
Started | 278 | 280
Completed (Data were locked on July 12, 2018 and were retrieved on August 14, 2018.) | 273 | 274
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Received Non-randomized Study Drug | 0 | 1
Not completed — Never Started Treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: The population analyzed is the Intention To Treat (ITT) Population, which included all participants who were randomized properly and who had received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oseltamivir | Placebo | Total
Number analyzed (Participants) | 277 | 279 | 556
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 271 | 273 | 544
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37 [27 to 49] | 35 [27 to 46] | 36 [27 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 164 | 347
  Male | 94 | 115 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 24
  Not Hispanic or Latino | 265 | 266 | 531
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 193 | 192 | 385
  Race: White | 74 | 76 | 150
  Race: Black or African American | 7 | 11 | 18
  Race: Race not available to clinic | 1 | 0 | 1
  Race: Subject does not know | 1 | 0 | 1
  Race: Subject does not want to report | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Argentina | 4 | 8 | 12
  United States | 91 | 87 | 178
  Thailand | 182 | 184 | 366
Confirmed influenza infection status by central testing [Count of Participants; unit: Participants] | 246 | 255 | 501
Influenza type/subtype by central testing [Count of Participants; unit: Participants]
  Influenza A/H3N2 | 122 | 129 | 251
  Influenza A/H1N1 | 39 | 54 | 93
  Influenza B | 85 | 71 | 156
  Negative | 30 | 22 | 52
  Co-infection | 0 | 1 | 1
  Missing | 1 | 2 | 3
Hours from onset of influenza-like illness to screening [Median (Full Range); unit: Hours] | 29 [1 to 49] | 27 [0 to 49] | 28 [0 to 49]
Hours from randomization to treatment initiation [Median (Full Range); unit: hours] | 1 [0 to 20] | 1 [0 to 21] | 1 [0 to 21]
Ever smoke tobacco [Count of Participants; unit: Participants] | 35 | 33 | 68
Vaccination for season of enrollment [Count of Participants; unit: Participants] | 34 | 23 | 57
BMI [Median (Inter-Quartile Range); unit: kg/m²] | 24.8 [22.1 to 29.3] | 24.7 [21.4 to 28.4] | 24.7 [21.6 to 28.7]
Overall symptom score, excluding 'other' [Median (Inter-Quartile Range); unit: units on a scale] — Symptoms were scored on a 4-point scale : 0=absent, 1=mild, 2=moderate, 3=severe.Overall symptom score was the sum of available scores for each of the 11 symptoms assessed (so ignoring missing values). The possible range of the overall symptom score is therefore 0 (no symptoms) to 33 (severe for all 11 symptoms). Subjects with missing evaluations for all symptoms were given a missing overall symptom score.
  units on a scale | 13 [10 to 17] | 13 [10 to 17] | 13 [10 to 17]
Global assessment in the morning at Day 0 [Count of Participants; unit: Participants]
  Subject feels as good today as before flu | 13 | 6 | 19
  Subject functions as well today as before flu | 49 | 40 | 89
Functional status [Median (Inter-Quartile Range); unit: units on a scale] — Average functional status was calculated as the average of the ten items assessed (so ignoring missing values), scoring 0='yes, limited a lot', 50='yes, limited a little', 100='no, not limited at all'. The possible range of the functional status score is therefore 0 (worst possible status) to 100 (best possible status). Subjects with missing evaluations for all items were coded as missing.
  units on a scale
    Pre-illness status | 100 [90 to 100] | 100 [95 to 100] | 100 [95 to 100]
    Day 0 status | 65 [40 to 75] | 65 [35 to 75] | 65 [40 to 75]
Complications of influenza [Count of Participants; unit: Participants]
  Sinusitis | 4 | 3 | 7
  Otitis Media | 0 | 1 | 1
  Bronchitis/Bronchiolitis | 4 | 2 | 6
  Pneumonia | 0 | 1 | 1
  Using antibiotic for other reasons | 6 | 5 | 11
Viral shedding by team-collected samples [Median (Inter-Quartile Range); unit: log10 copies/mL] — Population: restricted to subjects with confirmed influenza in a study team collected swab on Day 0
  log10 copies/mL
    number analyzed (Participants) | 246 | 255 | 501
    (all) | 6.9 [5.8 to 7.6] | 6.9 [5.9 to 7.6] | 6.9 [5.8 to 7.6]
Category of virus by team-collected samples [Count of Participants; unit: Participants] — LOD(limit of detection) /LLOQ(lower limit of quantification) for Influenza A and Influenza B by qPCR is 3.2/3.9 and 3.4/4.0, respectively.Results <LOD were imputed as LOD; results >=LOD and <LLOQ were imputed as LLOQ. Population: restricted to subjects with confirmed influenza in a study team collected swab on Day 0
  Participants
    number analyzed (Participants) | 246 | 255 | 501
    >= LLOQ | 237 | 245 | 482
    >= LOD, < LLOQ | 6 | 5 | 11
    < LOD | 3 | 5 | 8
Viral shedding by self-collected samples [Median (Inter-Quartile Range); unit: log10 copies/mL] — Population: restricted to subjects with confirmed influenza in a study team collected swab on Day 0
  log10 copies/mL
    number analyzed (Participants) | 246 | 255 | 501
    (all) | 6.1 [4.9 to 6.9] | 6.2 [5.4 to 6.9] | 6.2 [5.2 to 6.9]
Category of virus by self-collected samples [Count of Participants; unit: Participants] — LOD(limit of detection) /LLOQ(lower limit of quantification) for Influenza A and Influenza B by qPCR is 3.2/3.9 and 3.4/4.0, respectively. Population: restricted to subjects with confirmed influenza in a study team collected swab on Day 0
  Participants
    number analyzed (Participants) | 246 | 255 | 501
    >= LLOQ | 217 | 225 | 442
    >= LOD, < LLOQ | 11 | 6 | 17
    < LOD | 17 | 23 | 40
    Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Virus Detectable by Quantitative PCR (qPCR) in Nasopharyngeal (NP) Swabs at Day 3 -- Team Collected Samples
Description: The central laboratory performed a qualitative PCR test on the NP sample from Day 0 team collected swap in order to confirm influenza infection and to determine the influenza type and subtype. For participants with a positive influenza test result at Day 0 from this qualitative PCR testing, the laboratory then performed qPCR testing of subsequent samples to quantify viral shedding.
Time Frame: At Day 3
Population: The population analyzed was restricted to the 455 participants who had a confirmed positive test (from team collected sample) for influenza by qPCR in the central laboratory testing and were not in the pilot study for IRC004. 6 participants (3 in each arm) had missing endpoint samples so were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 220 | 229
Participants | 99 | 131
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; Assuming that pooled percentage of participants with virus detectable by PCR at Day 3 is 50%, assuming that the Oseltamivir arm was better than the placebo arm and that the detectable rate in the Oseltamivir arm was 42.5% compared to 57.5% in the placebo arm (a 15% reduction), and assuming 10% subjects with missing qPCR at Day 3, in a two-sided, two-sample 0.05-level t- test with 546 participants combined across both arms, there was 90% power; Test type: Superiority; p = 0.0097, Z-test, 2-sided — P-value was not adjusted for multiple interim analyses; Comparison of randomized arms was based on the normal approximation to the binomial distribution; Mean Difference (Final Values) = -12.2, 95% CI 2-sided [-21.4 to -3.0], Standard Error of Mean 4.6 — The difference in percents was calculated as the percent detectable in the Oseltamivir arm minus the percent detectable in the Placebo arm

2. Secondary Outcome: Number of Participants by Virus Detection Status--Team Collected Samples
Description: Number of participants who had undetectable values (less than the limit of detection [LOD]), who had values between the LOD and the lower limit of quantification (LLOQ), and who had values ≥LLOQ
Time Frame: At Day 0, 3 and 7
Population: The population analyzed is the Primary Efficacy Population (PEP), which included all participants who were randomized properly, had received at least one dose of study drug, and had influenza virus isolated and typed(from team collected sample) in the qualitative PCR evaluation at Day 0 from central laboratory testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 246 | 255
Participants
  Day 0: >= LLOQ | 237 | 245
  Day 0: >= LOD, < LLOQ | 6 | 5
  Day 0: < LOD | 3 | 5
  Day 0: Missing | 0 | 0
  Day 3: >= LLOQ | 85 | 109
  Day 3: >= LOD, < LLOQ | 24 | 36
  Day 3: < LOD | 134 | 107
  Day 3: Missing | 3 | 3
  Day 7: >= LLOQ | 16 | 21
  Day 7: >= LOD, < LLOQ | 11 | 5
  Day 7: < LOD | 214 | 224
  Day 7: Missing | 5 | 5

3. Secondary Outcome: qPCR Viral Shedding -- Team Collected Samples
Description: Median, 25% and 75% percentile of the value of viral shedding (Results <LOD were imputed as the LOD value, and Results >= LOD, <LLOQ were imputed as the LLOQ value.)
Time Frame: At Day 0, 3 and 7
Population: The population analyzed is the Primary Efficacy Population (PEP), which included all participants who were randomized properly, had received at least one dose of study drug, and had influenza virus isolated and typed (from team collected sample) in the qualitative PCR evaluation at Day 0 from central laboratory testing.
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 246 | 255
log10 copies/mL
  Day 0 | 6.85 [5.8 to 7.6] | 6.9 [5.9 to 7.6]
  Day 3 | 3.4 [3.2 to 4.5] | 3.9 [3.2 to 4.9]
  Day 7 | 3.2 [3.2 to 3.4] | 3.2 [3.2 to 3.4]

4. Secondary Outcome: Number Of Participants Shedding Virus -- Team Collected Samples
Description: Number of participants with undetectable viral load at both Day 3 and Day 7; detectable at Day 3 and undetectable at Day 7; detectable at Day 7 (irrespective of whether or not detectable at Day 3).
Time Frame: At day 3 and 7.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 246 | 255
Participants
  Undetectable at both Day 3 and 7 | 126 | 100
  Detectable at Day 3 and undetectable at Day 7 | 87 | 124
  Detectable at Day 7 | 27 | 26
  Missing result at Day 3 and/or Day 7 | 6 | 5
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; Test type: Superiority; p = 0.0243, Wilcoxon (Mann-Whitney) — P-value was not adjusted for multiple interim analyses

5. Secondary Outcome: Time to Alleviation of Influenza Clinical Symptoms
Description: The assessed symptoms were cough, nasal obstruction (stuffy nose), sore throat, fatigue, headache, muscle aches, feverishness, rhinorrhea, nausea, vomiting, diarrhea. Duration of clinical symptoms was defined as the time from Day 0 to the first of two successive measurements at which all clinical symptoms were grade 0 (absent) or 1 (mild). A measurement was considered to be the 8AM or 8PM assessment during Days 0 to 7 (so two measurements were obtained per day) and then the daily assessment thereafter. Time was calculated in half-days through to Day 7. If a subject's first two assessments on (baseline assessment and first subsequent diary card assessment) satisfied this criterion, then the duration was set to zero. For participants who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with symptoms evaluated.
Time Frame: From treatment initiation to Day 28
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 277 | 279
days | 4 [3.5 to 4.5] | 4 [3.5 to 4.5]
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; Test type: Superiority; p = 0.41, Log Rank — P-value was not adjusted for multiple interim analyses

6. Secondary Outcome: Time to Absence of Fever
Description: Fever was considered present based on the diary cards if a subject reported a maximal temperature ≥38.0°C (for the period since the diary card was previously completed) or reported having taken an antipyretic drug (also for the period since the diary card was previously completed). Otherwise, fever was considered not present during the period since the diary card was previously completed, except that the evaluation was considered missing if either the temperature or the antipyretic drug use entry was not completed on the diary card. The duration of fever was defined as the time from Day 0 to the first of two successive assessments (through to Day 7) or to the first assessment (Day 8 onwards) at which no fever was present according to this definition.For participants who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with fever evaluated.
Time Frame: From treatment initiation to Day 28
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 277 | 279
days | 1 [0.5 to 1.0] | 1 [0.5 to 1.0]
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; Test type: Superiority; p = 0.88, Log Rank — P-value was not adjusted for multiple interim analyses

7. Secondary Outcome: Time to Resolution of All Symptoms AND Fever
Description: The assessed symptoms were cough, nasal obstruction (stuffy nose), sore throat, fatigue, headache, muscle aches, feverishness, rhinorrhea, nausea, vomiting, diarrhea. Fever was considered present based on the diary cards if a subject reported a maximal temperature ≥38.0°C (for the period since the diary card was previously completed) or reported having taken an antipyretic drug (also for the period since the diary card was previously completed). Time to resolution of all clinical symptoms and fever is defined as the time from Day 0 to the first of two successive measurements at which all clinical symptoms are grade 0 (absent) or 1(mild) and no fever >=38.0 C or antipyretic drug is reported. For participants who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with symptoms and fever evaluated.
Time Frame: From treatment initiation to Day 28
Population: The population analyzed is the Intention To Treat (ITT) Population, which includes all participants who were randomized properly and who had received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 277 | 279
days | 4.0 [3.5 to 4.5] | 4.0 [3.5 to 4.5]
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; Test type: Superiority; p = 0.7461, Log Rank — P-value was not adjusted for multiple interim analyses

8. Secondary Outcome: Time to Feeling as Good as Before the Onset of the Influenza Illness
Description: Time to feeling as good as before influenza is defined as time to the first of two successive 'yes' responses to the question of 'feeling as good as you did before you had the flu'.For participants who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with question answered.
Time Frame: From treatment initiation to Day 28
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 277 | 279
days | 6.0 [5.0 to 6.5] | 6.0 [5.5 to 6.5]
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; Test type: Superiority; p = 0.1501, Log Rank — P-value was not adjusted for multiple interim analyses

9. Secondary Outcome: Time to Return to Pre-influenza Function
Description: Time to return to pre-influenza function is defined as the time from Day 0 to the first of two successive 'Yes' answers to the global assessment question 'Are you functioning as well as you were before you had the flu'.For participants who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with question answered.
Time Frame: From treatment initiation to Day 28
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 277 | 279
days | 3.5 [3.5 to 4.5] | 5.0 [4.0 to 5.0]
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; Test type: Superiority; p = 0.3025, Log Rank — P-value was not adjusted for multiple interim analyses

10. Secondary Outcome: Time to Return of Physical Function to Pre-illness Level
Description: Time to return of physical function to pre-illness level was defined as the time from Day 0 to the first of two successive measurements at which the physical function score equals or is better than the pre-illness score (obtained by recall at enrollment). For subjects who did not have two successive records meeting this criterion, follow-up was censored for analysis purposes at the time of the last but one diary card record with physical function evaluated.
Time Frame: From treatment initiation to Day 28
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 277 | 279
days | 7.0 [6.0 to 8.0] | 7.0 [6.0 to 7.0]
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; Test type: Superiority; p = 0.5466, Log Rank — P-value was not adjusted for multiple interim analyses

11. Secondary Outcome: Number of Participants With Treatment Compliance Status
Description: For each of the 5 days of treatment, participants were asked whether they took all study drug for that day. All participants were assumed to have taken at least some study drug even if they had zero days with all study drug reported as taken. Missing reports for some or all days were imputed as not having taken all study drug for the days concerned.
Time Frame: From treatment initiation to Day 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 277 | 279
Participants
  0 day with all study drug reported as taken | 1 | 2
  1 day with all study drug reported as taken | 2 | 2
  3 days with all study drug reported as taken | 2 | 1
  4 days with all study drug reported as taken | 2 | 1
  5 days with all study drug reported as taken | 270 | 273

12. Secondary Outcome: Percentage of Participants Who Required Hospitalization.
Description: The percentage of participants hospitalized by 28 days was constructed by inverting an exact binomial test of the actual percentages (ignoring loss to follow-up).
Time Frame: From treatment initiation to Day 28
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 277 | 279
percentage of participants | 1.4 [0.4 to 3.7] | 0.7 [0.1 to 2.6]
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; Test type: Superiority; p = 0.5311, two-sample binomial exact test — P-value was not adjusted for multiple interim analyses; The two-sample binomial exact test was performed in PROC STATXACT; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-1.4 to 3.0] — The difference in percents was calculated as the percent in the Oseltamivir arm minus the percent in the placebo arm

13. Secondary Outcome: Percentage of Participants Who Develop Bronchitis, Pneumonia, or Other Complications Requiring An Antibiotic Use, After Day 0.
Description: Participants were assessed for the signs/symptoms suggestive of one of the following complications: Sinusitis, Otitis Media ,Bronchitis / Bronchiolitis, Pneumonia and antibiotic use for reason other than above.
Time Frame: From treatment initiation to Day 28
Population: The population analyzed is the Intention To Treat (ITT) Population, which included all participants who were randomized properly and who had received at least one dose of study drug. The categories in the table are not mutually exclusive (because some participants had multiple complications) and the last row of the table summarizes all incidents.
Measure: Number; unit: percentage of participants
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 277 | 279
percentage of participants
  Sinusitis | 3.2 | 1.8
  Otitis Media | 0.4 | 0.4
  Bronchitis Bronchiolitis | 2.5 | 2.2
  Pneumonia | 0.4 | 0.4
  Antibiotic use | 2.5 | 3.6
  If have at least one Complication | 7.2 | 6.8
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; This test compared the difference in percentages of participants with at least one complication between two randomized arms; Test type: Superiority; p = 0.8498, Z test — P-value was not adjusted for multiple interim analyses; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-3.8 to 4.7] — The difference in percents was calculated as the percent in the Oseltamivir arm minus the percent in the placebo arm

14. Secondary Outcome: 28-day Mortality
Description: Number of deaths
Time Frame: From treatment initiation to Day 28
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 277 | 279
Participants | 0 | 0

15. Secondary Outcome: Percentage of Participants With Virus Detectable by Quantitative PCR (qPCR) in Nasopharyngeal (NP) Swabs --Self Collected Samples
Description: For participants with a positive influenza test result at Day 0 from qualitative PCR testing on the team collected sample, the laboratory then performed qPCR testing of self-collected samples to quantify viral shedding.
Time Frame: At Day 3
Population: The population analyzed was restricted to the 455 participants who had a confirmed positive test (from team collected sample) for influenza in the central laboratory testing and were not in the pilot study for IRC004. 9 participants (4 in the Oseltamivir arm and 5 in the Placebo arm) had missing endpoint samples so were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 219 | 227
Participants | 56 | 89
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; Test type: Superiority; p = 0.0021, Z test — P-value was not adjusted for multiple interim analyses; Mean Difference (Final Values) = -13.6, 95% CI 2-sided [-22.2 to -5.1]; The difference in percents was calculated as the percent with detectable in the Oseltamivir arm minus the percent with detectable in the placebo arm

16. Secondary Outcome: Number of Participants by Virus Detection Status --Self Collected Samples
Description: Number of participants who had undetectable values (less than the limit of detection [LOD]), who had values between the LOD and the lower limit of quantification (LLOQ), and who had values ≥LLOQ. Evening samples on Day 0, 1 and 2 were only required under protocol versions 1.0-4.0 and so were only collected for about 20% of participants.
Time Frame: At Day 0, Day 0 evening, Day 1, Day 1 evening, Day 2, Day 2 evening and Day 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 246 | 255
Participants
  Day 0: >= LLOQ | 217 | 225
  Day 0: >= LOD, < LLOQ | 11 | 6
  Day 0: < LOD | 17 | 23
  Day 0: Missing | 1 | 1
  Day 0 evening: >= LLOQ | 37 | 48
  Day 0 evening: >= LOD, < LLOQ | 4 | 1
  Day 0 evening: < LOD | 8 | 5
  Day 0 evening: Missing | 197 | 201
  Day 1: >= LLOQ | 138 | 147
  Day 1: >= LOD, < LLOQ | 30 | 27
  Day 1: < LOD | 75 | 76
  Day 1: Missing | 3 | 5
  Day 1 evening: >= LLOQ | 23 | 29
  Day 1 evening: >= LOD, < LLOQ | 4 | 9
  Day 1 evening: < LOD | 24 | 13
  Day 1 evening: Missing | 195 | 204
  Day 2: >= LLOQ | 70 | 92
  Day 2: >= LOD, < LLOQ | 26 | 31
  Day 2: < LOD | 146 | 129
  Day 2: Missing | 4 | 3
  Day 2 evening: >= LLOQ | 11 | 12
  Day 2 evening: >= LOD, < LLOQ | 6 | 4
  Day 2 evening: < LOD | 32 | 41
  Day 2 evening: Missing | 197 | 198
  Day 3: >= LLOQ | 39 | 65
  Day 3: >= LOD, < LLOQ | 25 | 35
  Day 3: < LOD | 178 | 149
  Day 3: Missing | 4 | 6

17. Secondary Outcome: qPCR Viral Shedding -- Self Collected Samples
Description: Median, 25% and 75% percentile of the value of viral shedding (Results <LOD were imputed as the LOD value, and Results >= LOD, <LLOQ were imputed as the LLOQ value.). Evening samples on Day 0, 1 and 2 were only required under protocol versions 1.0-4.0 and so were only collected for about 20% of participants.
Time Frame: At Day 0, Day 0 evening, Day 1, Day 1 evening, Day 2, Day 2 evening and Day 3
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 246 | 255
log10 copies/mL
  Day 0 | 6.1 [4.9 to 6.9] | 6.2 [5.4 to 6.9]
  Day 0 evening | 5.5 [4.3 to 6.2] | 6.0 [5.0 to 6.6]
  Day 1 | 4.2 [3.4 to 5.5] | 4.5 [3.4 to 5.9]
  Day 1 evening | 3.9 [3.2 to 7.2] | 4.0 [3.4 to 5.6]
  Day 2 | 3.4 [3.2 to 4.3] | 3.4 [3.2 to 4.8]
  Day 2 evening | 3.2 [3.2 to 3.9] | 3.2 [3.2 to 3.9]
  Day 3 | 3.2 [3.2 to 3.9] | 3.4 [3.2 to 4.0]

18. Secondary Outcome: Area Under The Curve (AUC) Of Viral Shedding For Self Collected Samples
Description: This AUC was calculated using the trapezoidal rule and the units of measurement are (days*log10 copies/mL) with the fact that it was the level of virus above the LLOQ being considered. The calculation of AUC was undertaken using measurements from Day 0 to Day 3 which were collected under all versions of the protocol (i.e. evening measurements on Days 0, 1 and 2 were not used as these were collected for only about 20% of subjects). Missing values during follow-up were ignored. This is equivalent to imputing a missing value using linear interpolation between the preceding and succeeding available values. For the five subjects with missing values following a last available measurement which was above the LLOQ, the remaining values were assumed to be the mean of preceding value and LLOQ in calculating the AUC.
Time Frame: From Day 0 to Day 3
Population: The population analyzed is the Primary Efficacy Population (PEP). The two subjects with missing values at Day 0 (one in each randomized arm) were excluded from this analysis.
Measure: Median (Inter-Quartile Range); unit: days*log10 copies/mL
Arm/Group | Oseltamivir | Placebo
Number analyzed (Participants) | 245 | 254
days*log10 copies/mL | 12.5 [11.35 to 14.55] | 13.18 [11.55 to 15.75]
Statistical Analysis 1: Comparison: Oseltamivir vs Placebo; Test type: Superiority; p = 0.022, Wilcoxon (Mann-Whitney) — P-value was not adjusted for multiple interim analyses

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the conduct of the study; from Day 0 to Day 28
Description: All worsening symptoms were evaluated as potential adverse events.If a diagnosis was clinically evident (or subsequently determined), the diagnosis, rather than the individual signs and symptoms or lab abnormalities, were recorded as the AE. All worsening laboratory values were also evaluated as potential adverse events. The DAIDS AE Grading Table (V1.0) was used.
Arm/Group | Oseltamivir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/277 | 0/279
Serious Adverse Events (participants affected / at risk) | 5/277 | 2/279
Other Adverse Events (participants affected / at risk) | 134/277 | 153/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir (N=277) | Placebo (N=279)
Influenza (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Chest pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oseltamivir (N=277) | Placebo (N=279)
Nausea (Gastrointestinal disorders) | 65 | 61
Diarrhoea (Gastrointestinal disorders) | 41 | 47
Vomiting (Gastrointestinal disorders) | 35 | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 32
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 | 25
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 26 | 23
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 20 | 16
Pyrexia (General disorders) | 31 | 27
Fatigue (General disorders) | 24 | 26
Headache (Nervous system disorders) | 28 | 24
Dizziness (Nervous system disorders) | 22 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 21
Hypertension (Vascular disorders) | 15 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT01314911/SAP_000.pdf
  • Study Protocol (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT01314911/Prot_001.pdf